CLINICAL TRIAL: NCT01818843
Title: Phase 1 Study of Inhaled Carbon Monoxide on the Effectiveness of Neonatal Pulmonary Hypertension
Brief Title: The Safety and Adverse Reaction Study of Neonatal to Inhaled Carbon Monoxide
Acronym: CO
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: CAN WANG (Other)
Collaborators: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Responsible Party: Sponsor-Investigator, CAN WANG, Phase 1 Study of Inhaled carbon monoxide on the effectiveness of neonatal pulmonary hypertension, Daping Hospital and the Research Institute of Surgery of the Third Military Medical University
Organization: Daping Hospital and the Research Institute of Surgery of the Third Military Medical University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DapingH 021
Record Dates: First submitted 2013-02-26; First posted 2013-03-27 (Estimated); Last update posted 2013-03-28 (Estimated); Status verified 2012-04

CONDITIONS: Miscellaneous Disorders in the Fetus or Newborn
Keywords: Carbon monoxide; safety; Adverse Reaction; newborn

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Safety and Adverse Reaction in CO (Experimental): Inhaled Carbon Monoxide
  Interventions: Other: Inhaled Carbon Monoxide

INTERVENTIONS:
Other: Inhaled Carbon Monoxide — Inhaled Carbon Monoxide in newborn

SUMMARY:
Based on the study about carbon monoxide in human inflammatory and other beneficial physiological function , now we'll be going to research its application in neonates .Phase 1 Study as a foundation for the further test is, the safety and Adverse reaction study of newborn to inhaled CO

DETAILED DESCRIPTION:
Previous studies have demonstrated that, carbon monoxide has showed the effectiveness such as in inflammation ,apoptosis as well as relaxation of smooth muscle of the body. Now we have a hypothesis to use carbon monoxide in pulmonary hypertension of the newborns, to observe whether it will decrease pulmonary artery hypertension on newborns. Phase 1 study is ,the safety and Adverse reaction study of newborn to inhaled CO , after this,we can master the application of carbon monoxide dose

ELIGIBILITY:
Inclusion Criteria:

* The newborn whose physiological function is healthy or close to healthy

Exclusion Criteria:

* Clinical considerations cannot survive or no treatment value of newborn Diagnosis of congenital or hereditary diseases, or children with heart diseaseCentral pulmonary vascular malformations in children

Ages: 1 Minute to 1 Month | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2012-04; Primary Completion 2013-01 (Actual); Study Completion 2013-12 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events | up to 1 month

CONTACTS AND LOCATIONS:
Locations (1):
- Daping Hospital, Chongqing, Chongqing Municipality, China